CLINICAL TRIAL: NCT01689103
Title: Therapeutic Alliances in Alcoholism Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Gerard J. Connors, Senior Research Scientist, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AA020253 (NIH)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Alcohol Use Disorders
Keywords: Alcohol use disorders; Treatment; Outpatient; Therapeutic alliance
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alliance Feedback to Therapist (Experimental): Alliance feedback provided to therapist
  Interventions: Behavioral: Cognitive-behavioral treatment
- No alliance feedback to therapist (Placebo Comparator): No alliance feedback provided to therapist
  Interventions: Behavioral: Cognitive-behavioral treatment

INTERVENTIONS:
Behavioral: Cognitive-behavioral treatment — Cognitive-behavioral treatment of alcohol use disorders
Behavioral: Cognitive-behavioral treatment — Cognitive-behavioral treatment for alcohol use disorders

SUMMARY:
This project is studying the role of the therapeutic alliance between the therapist and patient in the outpatient treatment of persons with alcohol use disorders.

DETAILED DESCRIPTION:
This project is studying the role of the therapeutic alliance between the therapist and patient in the outpatient treatment of persons with alcohol use disorders. Alliances are assessed over the course of treatment and will be reviewed in the context of posttreatment functioning.

ELIGIBILITY:
Inclusion Criteria:

* Current Alcohol Dependence diagnosis
* Live within commuting distance of treatment program
* Minimum 6th grade reading level
* Provide consent

Exclusion Criteria:

* Presence of current organic mental disorder, schizophrenia, or another psychotic disorder
* Treatment for an alcohol use disorder in past 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-08; Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent | 12 months

SECONDARY OUTCOMES:
Drinks per Drinking Day | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerard J Connors, Ph.D., Principal Investigator — University at Buffalo; Stephen A Maisto, PhD, Principal Investigator — Syracuse University; Ronda L Dearing, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Research Institute on Addictions, Buffalo, New York, United States

REFERENCES:
- [Derived] Rivera AP, Maisto SA, Connors GJ, Schlauch RC. Therapists' first impression of treatment motivation moderates the relationship between the client-rated therapeutic alliance and drinking outcomes during treatment. Alcohol Clin Exp Res (Hoboken). 2023 Apr;47(4):806-821. doi: 10.1111/acer.15040. Epub 2023 Mar 2. PMID 36863860